CLINICAL TRIAL: NCT05092165
Title: Methylene Blue for the Prevention of Hypotension During Hemodialysis: a Randomized Open Label Trial
Brief Title: Methylene Blue for the Prevention of Hypotension During Hemodialysis
Acronym: BLUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Chief of Critical Care Department, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLUE
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; Shock
MeSH Terms: conditions — Acute Kidney Injury; Shock | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene Blue (Active Comparator): Methylene blue will be infused during renal replacement therapy
  Interventions: Drug: Methylene Blue
- Control (Other): usual care
  Interventions: Other: Control

INTERVENTIONS:
Drug: Methylene Blue — 1 mg per kilogram bolus, followed by 0.1 milligram per kilogram during renal replacement therapy
  Arms: Methylene Blue
Other: Control — Usual care during renal replacement therapy
  Arms: Control

SUMMARY:
Hypotension is a common complication of intermittent renal replacement therapy. Methylene blue, an inhibitor of nitric oxide synthesis, has been suggested to improve hemodynamics during renal replacement therapy in ambulatory patients, but evidence is lacking for critically ill patients.

This trial will assess whether methylene blue can improve hemodynamics and blood pressure for patients with shock requiring renal replacement therapy.

DETAILED DESCRIPTION:
This is a single-center, randomized, non-blind study, with a intention-to-treat analysis, aiming to evaluate whether the use of methylene blue reduces the incidence of hypotension during hemodialysis, resulting in a reduction in the need for therapeutic modifications during the session, defined as interruption session, reduced fluid losses and increased need for vasopressors. Patients will be randomized using RedCap platform in variable blocks of 4-6, stratified by center in a 1:1 ratio and by previous use of vasopressors, into two groups, intervention and usual treatment. Access to randomization will be available 24 hours, 7 days a week. Patients on intermittent renal replacement therapy will be selected to receive or not methylene blue at a bolus dose of 1 mg/kg, followed by a continuous infusion of 0.1 mg/kg of body weight in a total of 200 ml of solution. saline throughout the dialysis session. The usual care group will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative accepted trial enrollment
2. Age above 18 years
3. Chronic or acute kidney injury in need for renal replacement therapy
4. Blood pressure lower than 100 mmHg or in use of any vasopressor

Exclusion Criteria:

1. Pregnancy
2. Death considered imminent in the next 24 hours
3. Patients not on full code status
4. Hypertensive patients where dialysis was indicated to remove fluids
5. Known allergy to methylene blue
6. Known glucose-6-phosphate deficiency
7. Previously enrolled in the trial
8. Acute coronary Syndrome
9. Domiciliary nitrate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint | 6 hours
  Composite endpoint of: Increase in vasopressor dose in at least 15% of initial dose or interruption of dialysis or reduction in ultrafiltration rate

SECONDARY OUTCOMES:
Hypotension | 6 hours
  Mean blood pressure below 65 mmHg for at least 5 minutes during renal replacement therapy
Maximum vasopressor dose | 24 hours
  Maximum vasopressor dose, in micro-grams per kilogram per minute used during de first 24 hours
Mortality in the intensive care unit | 60 days
  Death in the intensive care unit
Mortality in the hospital | 60 days
  Death during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Carla Pontes, MD, Principal Investigator — Federal University of São Paulo; Flavia R Machado, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after trial is published
Access Criteria: After aproval by the executive comittee